CLINICAL TRIAL: NCT05910606
Title: Strong Foundations 2.0: A Digitally Delivered Fall Prevention Program for Remote Deployment of Exercise in an At-risk Population of Older Adults.
Brief Title: Strong Foundations 2.0: A Digitally Delivered Fall Prevention Program.
Acronym: SF2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ryan Moran, Associate Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 806696
Record Dates: First submitted 2023-05-24; First posted 2023-06-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Fall Prevention; Bone Health; Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Experimental): Digitally delivered strength, balance and postural control exercises
  Interventions: Behavioral: Digital Exercise

INTERVENTIONS:
Behavioral: Digital Exercise — Fall Prevention Program: Our fall- risk reduction program overs digitally delivered exercise with real time feedback from expert instructors.

SUMMARY:
Study Description: The investigators propose to extend earlier research conducted during a feasibility study (Strong Foundations 1.0) by enrolling participants who have a greater risk for falling (x4 cohorts of up to 15 individuals) and from a lower socio-economic status (x4 cohorts of up to 15 individuals), and by collecting high quality laboratory based measures of balance, posture, and strength to better determine the effectiveness of the program and its suitability for widespread deployment.

Additionally, the investigators hope to showcase it is feasible to sustain programmatic gains with ongoing digitally delivered content by combining cohorts into a larger group that continues to practice the foundational exercises taught during the 12-week initial program.

DETAILED DESCRIPTION:
Study Description: The investigators have successfully completed a pilot project focused on feasibility and user acceptability of a digitally delivered program for fall prevention in older adults. This program was well received among participants of lower risk individuals, and with this extension we will be exploring the acceptability, utility, and scalability in both a higher risk and lower socio-economic status group of older adults.

The primary goal of this program is to reduce fall risk using a digitally delivered exercise intervention with a high level of personalized instruction for the initial portion of the intervention (12 weeks) and to maintain any established reduction in fall risk in an ongoing, pooled cohort extended beyond the initial 12 weeks of training that features a smaller amount of personalized instruction .

The investigators will extend earlier research using a digitally delivered fall-prevention exercise program by engaging 1) two cohorts of up to 15 individuals each at low to average risk of falls and 2) two additional cohorts, of up to 15 individuals with established risk factors for falling identified from the larger San Diego community and a similar number of cohorts/individuals in collaboration with community partners who provide housing for a population from lower socio-economic status, and potentially less access to, and comfort with digital technology. Thus, in total the investigators will enroll up to 120 participants across all sites/settings through this timeframe.

Description of Study Intervention:

Strong Foundations is a 12 week iterative curricular program with three core components: postural alignment and control, balance and mobility, and muscular strength and power. All the exercises offered over the course of the intervention are appropriate for the target population and are standardized so all participants receive the same basic instruction, but level of difficulty is scaled to participant experience, capability, and musculoskeletal limitations.

This fall- risk reduction program, Strong Foundations was designed to be delivered digitally, and while there are many such programs currently available on the internet, especially in the time of COVID-19, the novel feature of this program is the delivery of semi-individualized instruction in real time within a small group setting. This is accomplished largely by use of the 'breakout room' feature on the Zoom platform, where 2-3 trained intern instructors correct form while the lead instructor teaches the larger group. The program was designed with physician input and by exercise physiologists and a Doctor of Physical Therapy candidate, all with extensive training in both group and individualized exercise for geriatric populations.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older, ambulatory, including with the use of a cane or walker, and able to read and speak English.
* Completion of the STEADI Stay Independent Questionnaire (with score of 6 or less)
* Access to internet/computer and Zoom-interface / broadband with a device with a minimum screen size of 7 inches (i.e. tablet or larger).

Exclusion Criteria:

* Individuals who are wheel-chair bound
* Score 7 or more on the STEADI modified questionnaire

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-07-16 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in the scores from the Short Physical Performance Battery (Balance) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Change in composite score and individual scores for all components Summary Score 0-12 with higher values being indicative of better performance. Positive change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention.
  Gait Speed: Measured in m/sec with higher values being indicative of better performance and lower risk Positive change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention 5 repetition chair stands: Scored in seconds with lower values being indicative of better performance and lower risk. Negative change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention Balance: 0-10 seconds with higher time indicative of better balance and lower risk. Positive change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention
Change in time to complete the Timed Up and Go (Balance and Function) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Change in the time to complete a standardized assessment of functional mobility and fall risk that times a participant's ability to get up out of chair, walk 8 feet, navigate an obstacle and return to a seated position
  Measured in seconds with variable possible length. Faster times are indicative of better performance and lower risk. Negative change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention
Change in postural sway during the Better Balance Testing (Balance) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Changes in the amount of movement (postural sway) observed during a standardized measure of balance on a force platform. This is a well validated measure of proprioceptive and vestibular function utilizing computerized dynamic posturography (i.e. balance board that measures center of pressure and postural sway)
  Measured in mm of sway with range 0 - ?. Lower scores are indicative of greater stability and lower risk. Negative change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention
Change in time to complete a 25 foot walk (Balance and function) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Change in time to complete a standardized assessment of gait speed and variability commonly used to assess fall risk.
  Measured in seconds to calculate gait speed in m/sec. Lower times (in sec) and higher speeds (in m/sec) are indicative of better function and lower risk. Negative change scores (T2-BL or T1-BL or T2-T1) for time will be associated with improved performance following intervention
Change in distance covered during a 2.5 minute walk (Aerobic Capacity) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Change in the distance (and estimated aerobic capacity derived from distance) on a standardized walk test to measure aerobic endurance and estimate overall capacity
  Measured in meters with variable range. Higher scores are indicative of greater cardiovascular function and lower risk. Positive change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention
Change in Grip Strength (Muscular Strength) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Change in a Standardized assessment to assess muscular strength. Used because it correlates well with overall body strength.
  Measured in kg for both hands and averaged with a variable range. Higher scores are indicative of greater muscular strength and lower risk. Positive change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention
Change in number of chair stands completed in 30 seconds (Muscular Strength) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Change in a common field measure associated with fall risk. Used to measure leg strength and endurance specifically.
Change in the amount of force generated during isometric assessment of leg strength using BIODEX System 4 PRO (Muscular Strength) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Change in the amount of force generated during maximal exertion for short time against an immovable object at 3 joint angles to measure hamstring and quadricep strength
Change in amount of force generated during isometric assessment of back strength using BIODEX System 4 PRO (Muscular Strength) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Chage in the amount of force generated during maximal exertion for short time against an immovable object at 3 joint angles to measure strength of the muscles surrounding the lumbar and thoracic spine. Positive change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention
Change in Occipital to Wall Distance (Posture) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Change in common measurement of the curvature of the thoracic and cervical spine done in standing position
  Score range is in mm and is variable. Higher values indicate more kyphotic curve and are associated with worse outcomes. Negative change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention
Change in the number of blocks used for the blocks measurement of Kyphosis (Posture) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Measurement of the curvature of the thoracic and cervical spine done in a supine position
  Range 0-7 with higher values indicative of more kyphosis and worse outcomes. Negative change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention
Change in height using multiple measures of height (Posture) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Changes in the difference between height measured while standing "normally" vs. "as tall as possible" to measure height loss due to spinal curvature in the absence of muscular engagement.
  Measurement in mm of difference with higher scores indicative of greater non specific postural imbalance/deformity and are associated with worse outcomes. Negative change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention
Change in hip Tilt and Shift (Posture) | Baseline, 12 weeks (post intervention), 24 weeks (post follow up)
  Changes in standardized physical therapy based assessments of left/right and forward/backward symmetry of hips, shoulders and ankles
  Measured in degrees with a likely range of 0-15. Greater values are indicative of non specific postural imbalance/deformity and are associated with worse outcomes. Negative change scores (T2-BL or T1-BL or T2-T1) will be associated with improved performance following intervention

SECONDARY OUTCOMES:
System Usability Scale | 12 weeks (post intervention)
  Validated Scale to assess program's accessibility and perceived usefulness. Score range 20-100 with higher scores being indicative of more perceived usability (i.e. greater acceptability)
User Experience | 12 weeks (post intervention)
  Non-standardized Likert scale questions asking about participant's experience with the digital format including feelings of safety, engagement, and program enjoyment. Range 1-5. Some are positively coded so that higher scores are indicative of better acceptability and some are negatively coded so that lower scores are indicative of better acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Health, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual data